CLINICAL TRIAL: NCT06621251
Title: Phase 2 Study to Evaluate the Efficacy and Safety of TRL1068 for the Treatment of Chronic Prosthetic Joint Infection of the Knee or Hip Without Exchange Arthroplasty
Brief Title: Study to Evaluate the Efficacy and Safety of TRL1068 for the Treatment of Prosthetic Joint Infection
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Trellis Bioscience LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRL1068-201
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Prosthetic Joint Infections of Hip; Prosthetic Joint Infections of Knee
Keywords: biofilm; antibiotic-resistant infections
MeSH Terms: interventions — TRL1068; Debridement; Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TRL1068 + DAIR (Experimental): TRL1068 will be administered at 15 mg/kg IV on Day 1 and subsequently at 7.5 mg/kg on Days 15, 29, and 43. Between Day 15-22, a DAIR procedure will be completed.
  Interventions: Drug: TRL1068 (calpurbatug), a human monoclonal antibody; Procedure: DAIR
- SoC (No Intervention): Standard of Care arm, receiving 2-stage surgery as is SoC for PJI. Reduced assessments will be done at the same timepoints as the experimental arm.

INTERVENTIONS:
Drug: TRL1068 (calpurbatug), a human monoclonal antibody — A human IgG1κ (G1m1,17 (z,a); Km3 allotype) monoclonal antibody
  Arms: TRL1068 + DAIR
Procedure: DAIR — DAIR procedure will be performed between days 15-22
  Other Names: debridement, antibiotics, and implant retention
  Arms: TRL1068 + DAIR

SUMMARY:
TRL1068 is expected to eliminate the pathogen-protecting biofilm in the prosthetic joint and surrounding tissue, thus making pathogens substantially more susceptible to established antibiotic treatment regimens. This Phase 2 study is designed to assess efficacy and safety of TRL1068 in combination with a DAIR (debridement, antibiotics, and implant retention) procedure for chronic prosthetic joint infections of the knee and hip, specifically, eliminating the need for the standard of care 2-stage exchange surgery, so that the original prosthesis can be retained.

DETAILED DESCRIPTION:
Approximately 75% of all clinically significant human infections are estimated to be biofilm-related. Prosthetic joint infections are a classical example of difficult to eradicate infections associated with biofilm. Most Prosthetic Joint Infection (PJI) cases are caused by staphylococcal species (~70%) with an increasing number being antibiotic-resistant (MRSA). In the US, two-stage revision is the standard of care for replacement of an infected prosthetic joint, and is associated with substantial costs and prolonged immobility. TRL1068 is a fully human antibody that has been shown in pre-clinical studies and in the first-in-human Phase 1 study TRL1068-101 to disrupt biofilm. TRL1068 targets a highly conserved epitope on the DNABII family of bacterial DNA binding proteins that includes histone-like (HU) and integration host factor (IHF) proteins of clinically relevant Gram-positive and Gram-negative bacteria. The DNABII epitope bound by TRL1068 has no homologs in the human proteome.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 85 years, inclusive
2. Chronic PJI:

   1. Systemic Host Grade of A or B [McPherson 2011] (Appendix 3) and either
   2. First chronic PJI of the hip or knee, confirmed by synovial fluid aspirate culture or
   3. Recurrent chronic PJI of the hip or knee confirmed by synovial fluid aspirate culture
3. Willing to be randomized to either:

   1. Receive TRL1068 and to be scheduled for DAIR between Day 15 + 7 days (i.e., between days 15-22) and 10 weeks of targeted antibiotic treatment or
   2. Participate in an observational study arm that receives SoC (i.e., two-stage prosthetic joint replacement) and

   i. Sonication of the explanted prosthesis and performance of synovial fluid aspirates ii. Consents to conduct of stage 2 (implantation of new prosthesis)
4. At least 1 positive bacterial culture without concomitant fungal infection from the infected joint (a joint aspirate within 28 days prior to Screening is acceptable)
5. All identified pathogen(s) are susceptible to the planned antibiotic regimen
6. Availability of radiology assessments of the affected joint without signs of loosening of the prosthesis or presence of osteomyelitis
7. Willing and able to provide written informed consent
8. Willing to perform and comply with all study procedures, including attending clinic visits as scheduled
9. Men and women of childbearing potential (WOCBP) must be willing to practice a highly effective method of contraception that may include, but is not limited to, abstinence, sex only with persons of the same sex, monogamous relationship with vasectomized partner, vasectomy, hysterectomy, bilateral tubal ligation, licensed hormonal methods, intrauterine device (IUD), or use of spermicide combined with a barrier method (e.g., condom, diaphragm) through Day 365.

Exclusion Criteria:

1. PJI associated with presence of concomitant fungal infection or bacterial pathogens that, even when in planktonic form (i.e., when released from biofilm), cannot be adequately treated with available antibiotics.
2. More than one draining sinus and single draining sinus of > 1 cm
3. Less than 3 years life expectancy based on underlying morbidities
4. Expected to receive chronic suppressive antibiotic therapy
5. Congestive heart failure; New York Heart Association (NYHA) Functional Classification of Heart Failure Grade > 3B
6. Uncontrolled diabetes, defined as hemoglobin A1c > 7.4%.
7. BMI > 45
8. Any acute illness within 14 days of Day 1 that could confound the evaluation of safety evaluation of TRL1068, especially local or systemic fungal and other known or suspected bacterial infections
9. Receiving or recently received another investigational drug (within 30 days of Day 1, or 5 half-lives of the investigational drug, whichever is longer)
10. Received any vaccine within 14 days prior to Day 1
11. Positive serum pregnancy test for WOCBP, or nursing women
12. History of drug or alcohol abuse that, in the opinion of the Investigator, would interfere with the patient's ability to comply with all study requirements
13. Any other comorbidity or condition that, in the opinion of the Investigator would make the patient unsuitable for the study or unable to comply with the study requirements.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy of TRL1068 in eliminating the need for an SoC 2-stage exchange arthroplasty | Day 365
  Incidence of resolved PJI, i.e., completion of planned surgical interventions for PJI (DAIR or 2-stage exchange arthroplasty), and not receiving systemic antibiotics for PJI or antibiotic suppression therapy for PJI or any other planned interventions to treat PJI by end of study.

SECONDARY OUTCOMES:
Duration (days) with resolved PJI | Day 365
  Days after completion of planned surgical interventions for PJI (DAIR or 2-stage exchange arthroplasty) without receiving systemic antibiotics for PJI or antibiotic suppression therapy of PJI or any other planned interventions to treat PJI by end of study.
Incidence of recurrent PJI across treatment groups | Day 365
  Recurrent PJI will include PJI in which the causative pathogen of the recurrent PJI was not identified at baseline.
Incidence of PJI reinfection across treatment groups | Day 365
Incidence, duration and severity of AEs or SAEs of secondary infections | Day 365
Musculoskeletal Infection Society (MSIS) Scores | Day 365
  MSIS scores on Day 1, day of DAIR (Day 15 + 7 days) versus Day 1, day of first stage of SoC and EOS (Day 365) that are indicative of the presence of PJI. MSIS Minor Criteria score range is 0-12, above or equal to 6 is infected, 2-5 is possibly infected, 0-1 is not infected.
Quality of life PROMIS-PF Short Form 6b | Day 365
  Quality of life as measured by the Quality of Life (QoL) Questionnaire (PROMIS-PF Short Form 6b). Score range is 6-30, with higher scores indicating higher functioning.
Resource utilization: duration of hospitalization as a result of PJI, SoC or surgical wound infection | Day 365
Resource utilization: need to stay in a rehabilitation center or other institution, e.g., nursing home as a result of PJI, SoC or surgical wound infection | Day 365
Incidence, duration and severity of AEs and SAEs across treatment groups | Day 365
  abnormal vital signs and safety labs will be documented as adverse events.

OTHER OUTCOMES:
Immunogenicity of TRL1068 as measured by anti-drug antibodies (ADAs) | Day 365
  The exploratory objective is to assess the immunogenicity of TRL1068 as measured by anti-drug antibodies (ADAs).
Pharmacokinetics - serum and synovial concentrations of TRL1068 | Day 365
  Serum and synovial concentrations of TRL1068 will be determined by ELISA
Pharmacodynamics - inflammatory biomarkers - CRP | Day 365
  CRP will be compared within and across groups
Pharmacodynamics - inflammatory biomarkers - ESR | Day 365
  ESR will be compared within and across groups

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - OrthoArizona, Gilbert, Arizona
  - University of Arkansas for Medical Sciences (UAMS), Little Rock, Arkansas
  - UCLA, Los Angeles, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Gulfcoast Research Institute, Sarasota, Florida
  - Phoenix Clinical Research, Tamarac, Florida
  - Sinai Hospital Baltimore, Baltimore, Maryland
  - New England Baptist Hospital, Boston, Massachusetts
  - NYU Langone Health, New York, New York
  - University of Rochester, Rochester, New York
  - M3 Wake Research Associates, Wilmington, North Carolina
  - Proactive RGV, Brownsville, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Houston Methodist, Houston, Texas
  - Paradigm Research Center, Houston, Texas
  - North Texas Medical Research Institute, Rockwall, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
The study results will be published after the study is completed.

REFERENCES:
- [Result] Conway J, Delanois RE, Mont MA, Stavrakis A, McPherson E, Stolarski E, Incavo S, Oakes D, Salvagno R, Adams JS, Kisch-Hancock A, Tenorio E, Leighton A, Ryser S, Kauvar LM, Bernthal NM. Phase 1 study of the pharmacokinetics and clinical proof-of-concept activity of a biofilm-disrupting human monoclonal antibody in patients with chronic prosthetic joint infection of the knee or hip. Antimicrob Agents Chemother. 2024 Aug 7;68(8):e0065524. doi: 10.1128/aac.00655-24. Epub 2024 Jul 16. PMID 39012102